CLINICAL TRIAL: NCT00135629
Title: Factors Predicting Efficacy of Allergen Injection Immunotherapy for Grass Pollen Hayfever: A Pilot Study. (Up-dosing Study)
Brief Title: Factors Predicting Efficacy of Allergen Injection Immunotherapy for Grass Pollen Hayfever
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Imperial College London (Other)
Collaborators: ALK-Abelló A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DHRG-UpDosing
Record Dates: First submitted 2005-08-25; First posted 2005-08-26 (Estimated); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Rhinitis, Allergic, Seasonal
Keywords: Hayfever; Sublingual Immunotherapy; Grass pollen immunotherapy; Late cutaneous response; Intradermal allergen challenge; Seasonal Allergic Rhinoconjunctivitis
MeSH Terms: conditions — Rhinitis, Allergic, Seasonal | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: 2 arm, randomized, double-blind trial
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunotherpy Arm (Experimental): 12 patients received active injections of an alum-adsorbed grass pollen vaccine
  Interventions: Biological: Active injections of alum-adsorbed grass pollen vaccine (Alutard SQ).; Procedure: Venepuncture: 100ml blood sample taken on 12 separate visits
- Placebo Arm (Placebo Comparator): 6 patients received placebo injections
  Interventions: Other: Placebo Injection; Procedure: Venepuncture: 100ml blood sample taken on 12 separate visits

INTERVENTIONS:
Biological: Active injections of alum-adsorbed grass pollen vaccine (Alutard SQ). — Active injections of alum-adsorbed grass pollen vaccine (Alutard SQ).
  Arms: Immunotherpy Arm
Other: Placebo Injection — Placebo Injection
  Arms: Placebo Arm
Procedure: Venepuncture: 100ml blood sample taken on 12 separate visits — Venepuncture: 100ml blood sample taken on 12 separate visits

SUMMARY:
The purpose of this study is to determine at which point in the dosing regime grass pollen immunotherapy causes a significant reduction in the late skin response to allergen challenge. A once weekly cluster regimen of 2 injections per visit was employed during the up-dosing phase, followed by monthly maintenance injections of 100,000 SQ units. Symptom scores and need of rescue medication were recorded by patients during the study period. The size of early and late cutaneous response to allergen challenge was recorded and measured by a physician.

DETAILED DESCRIPTION:
This was a single centre, randomised, double-blind placebo controlled trial of grass pollen injection immunotherapy (Alutard SQ, ALK Abello, Denmark) in adults with severe summer hayfever unresponsive to antihistamines and topical steroids. The main aim was to determine at which point in the dosing regime grass pollen immunotherapy causes a significant reduction in the late skin response to allergen challenge. A once weekly cluster regimen of 2 injections per visit was employed during the up-dosing phase, followed by monthly maintenance injections of 100,000 SQ units. Twelve patients received active treatment (mean age 31, 7 male) whilst 6 were given placebo (mean age 37, 2 male). The 24 hour skin response (size of swelling, (mm)) to intradermal allergen challenge (0.1, 1, 10 BU) was determined on alternate weeks during the 8 week up-dosing phase and then monthly up to 6 months and 3 monthly up to 11-13 months following initiation of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male and female 18-65 years of age
* Written informed consent obtained before entering the trial
* A clinical history of grass pollen induced allergic rhinoconjunctivitis of two years or more requiring treatment during the grass pollen season
* A clinical history of severe rhinoconjunctivitis symptoms (interfering with usual daily activities or sleep), which remain troublesome despite treatment with anti-allergic drugs during the grass pollen season
* Positive Skin Prick Test (SPT) response (wheal diameter ≥ 3 mm) to Phleum pratense
* Positive specific IgE against Phleum pratense (≥ IgE Class 2)
* Physical examination with no clinically relevant findings
* If pre-menopausal female of childbearing potential, the subject must test negative on standard urine pregnancy test and must be willing to practice appropriate contraceptive methods for the duration of the trial
* Willingness to comply with this protocol

Exclusion Criteria:

* FEV1 < 70% of predicted value
* A clinical history of symptomatic seasonal allergic rhinitis and/or asthma due to tree pollen or weed pollen adjacent to the start of - and potentially overlapping - the grass pollen season
* A clinical history of significant symptomatic perennial allergic rhinitis and/or asthma caused by an allergen to which the subject is regularly exposed
* A clinical history of significant recurrent acute sinusitis (defined as 2 episodes per year for the last two years all of which required antibiotic treatment) or chronic sinusitis
* At randomisation, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media or other relevant infectious process (serous otitis media is not an exclusion criterion)
* History of emergency visit or admission for asthma in the previous 12 months
* Use of an investigational drug within 30 days prior to screening
* Previous treatment by immunotherapy with grass pollen allergen or any other allergen within the previous 5 years
* History of anaphylaxis, including anaphylactic food allergy, bee venom anaphylaxis, exercise anaphylaxis or drug induced anaphylaxis
* History of angioedema
* Any of the following underlying conditions known or suspected to be present:

  * Cystic fibrosis
  * Malignancy
  * Insulin-dependent diabetes
  * Malabsorption or malnutrition
  * Renal or hepatic insufficiency
  * Chronic infection
  * Drug dependency or alcoholism
  * Ischemic heart disease or angina requiring current daily medication or with any evidence of disease making implementation of the protocol or interpretation of the protocol results difficult or jeopardising the safety of the subject (e.g. clinically significant cardiovascular, serious immunopathologic, immunodeficiency whether acquired or not, hepatic, neurologic, psychiatric, endocrine, or other major systemic disease)
* Immunosuppressive treatment
* History of hypersensitivity to the excipients of the trial medications
* History of allergy, hypersensitivity or intolerance to trial medications or rescue medications
* A mental condition rendering the subject unable to understand the nature, scope and possible consequences of the trial, and/or evidence of an uncooperative attitude
* Unlikely to be able to complete the trial, for any reason, or likely to travel for extended periods of time during the grass pollen season

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2002-10; Primary Completion 2008-01 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Symptom and medication score recorded by subjects | Assessment scores obtained after 12 months of treatment
  Overall assessment of symptoms was recorded on a numeric scale (-3 to +3) by each patient at the end of the study
Adverse events (conjunctival symptoms) | 10 minutes post-conjunctival allergen provocation after 12 months of treatment
  Conjunctival symptoms elicitation with P-pratense allergen (reduced response detection)

SECONDARY OUTCOMES:
Intradermal allergen challenge | Biweekly during up-dosing and then monthly upto 6 months, and up to 12 months following initiation of treatment.
  All patients underwent re-peated venesection and intradermal allergen challenge for testing of early and late skin responses: allergen-induced cytokine production over 10 months (reduced response change to P pratense-specific antigens). Intradermal allergen challenge for testing of early and late skin responses at biweekly intervals during updosing and at monthly intervals during the maintenance phase.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen R Durham, Professor, Principal Investigator — Royal Brompton Hospital, Imperial College, National Heart & Lung Institute
Locations (1):
- Royal Brompton Hospital, NHLI Imperial College, London, United Kingdom

REFERENCES:
- [Result] Francis JN, James LK, Paraskevopoulos G, Wong C, Calderon MA, Durham SR, Till SJ. Grass pollen immunotherapy: IL-10 induction and suppression of late responses precedes IgG4 inhibitory antibody activity. J Allergy Clin Immunol. 2008 May;121(5):1120-1125.e2. doi: 10.1016/j.jaci.2008.01.072. Epub 2008 Apr 18. PMID 18374405